CLINICAL TRIAL: NCT06634537
Title: Effect of Hard and Soft Density Insoles on the Postural Control of Adults Over 65 Years of Age
Brief Title: Effect of Insoles on the Postural Control of Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Vicenta Martínez Córcoles, Principal Investigator PhD, Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23/604-E
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postural; Defect; Adult; Orthopedic
Keywords: BALANCE; insoles; barefoot; olders adults

STUDY DESIGN:
Intervention Model Description: Longitudinal
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Comparator: Insoles soft and hard and barefoot (Experimental): Experimental: Active Comparator: Insoles soft The pattern will be performed 3 times per day (10 repetitions, 30 seconds each repetition). A daily Active Comparator: Insoles hard and barefoot en 3 month and 6 month.
  Interventions: Device: Active Comparator: insoles hard, soft and barefoot
- Active Comparator: Insoles hard and soft and barefoot (Experimental): Experimental: Active Comparator: Insoles hard The pattern will be performed 3 times per day (10 repetitions, 30 seconds each repetition). A daily Active Comparator: Insoles hard and barefoot en 3 month and 6 month.
  Interventions: Device: Active Comparator: insoles hard, soft and barefoot
- Active Comparator: barefoot and insoles hard and soft (Experimental): Experimental: Active Comparator: barefoot The pattern will be performed 3 times per day (10 repetitions, 30 seconds each repetition). A daily Active Comparator: Insoles hard and barefoot en 3 month and 6 month.
  Interventions: Device: Active Comparator: insoles hard, soft and barefoot

INTERVENTIONS:
Device: Active Comparator: insoles hard, soft and barefoot — Primary Outcome Measure:
  1. Stabilometry The measurements were conducted University. To assess participants' balance, the anthropometric position of the protocol proposed by the International Society for the Advancement of Cineatropometry (ISAK) was assigned: participants placed their mi Frankfort; the upper limbs remained relaxed throughout the body, with palms facing forward and thumbs separated from the rest of the toes, and were barefoot with feet externally rotated f 30 degrees and with a heel distance of 4cm.
  The children were wearing sports costumes to contribute their free movement. For stabilometry data collection will use an inertial measurement instrument called Gyko® It is a state-of-the-art device that allows to measure an objective assessment of acceleration, angular velocity and with an acquisition frequency of 100Hz [Time Frame: pre intervention, 3 months post intervention, 6 months post intervention]
  Other Names: Effet in postural control of hard and soft density insoles

SUMMARY:
Background: there is a high risk of falls in older adults. One of the factors contributing to fall episodes is advancing age due to deterioration of the proprioceptive system. Certain clinical procedures improve balance and posture such as the use of insoles.

Objetive: to evaluate the impact of hard and soft insoles on static foot balance in healthy older adults compared to barefoot people.

Methods: a clinical trial was conducted with a sample size of 31 healthy with a mean age of 69.03±3.82 years. Postural control willevaluated in different conditions of barefoot balance with hard and soft insoles.

DETAILED DESCRIPTION:
All subjects completed three testing sessions in a laboratory setting without external distraction. The same testing procedures were repeated during each session, with a time period of one week between sessions. All participants were asked for their information (age, sex, weight, height and date of birth), and they were then asked to take off their shoes in order to take the measurements. The Gyko® device was then placed in a harness on the back of the participant, who was subsequently asked to remain in an anthropometric position.

During the first testing session, postural impacts were assessed whilst subjects will barefoot. In the second testing session, subjects wore a soft gel insole: Cushioning gel slim (SIDAS, 18, rue Léon Béridot, Voiron, France: https://www.sidas.com/es/plantillas-para-el-uso-diario/156-cushioning-gel.html). During the third and final test, Winter+ insoles were used (SIDAS, 18, rue Léon Béridot, Voiron, France; https://www.sidas.com/es/plantillas-esqui-snowboard/221-winter-plus.html) .

Each session lasted around 30 seconds, data will collected while standing, with participants in in a bilateral stance. Each task was performed both with eyes open and eyes closed. To control for possible variations in visual field, subjects were asked to focus on a target placed 2 meters in front of them at eye level. If the person moved or lost balance, the data was discarded and the test was repeated until it was obtained correctly.

In each test, the data was managed as follows; the first 10 seconds of each test were discarded; the average of the remaining 20 seconds was taken for later analysis. Postural sway was assessed using a set of measures. The sway area (cm2) will calculated using the area of the ellipse generated by the software. Additionally, sway distance and sway velocity were assessed along the anterior-posterior and medial-lateral axes

ELIGIBILITY:
Inclusion Criteria:

* The insoles involved are standard insoles which are not used to correct deformities; the differences between them concern the density of the materials (higher density is harder and lower density is softer). Participants could have any existing foot condition or deformity.
* Each pre-existing foot condition or deformity would be noted and listed for the sole purpose of evaluating the relationship between postural control and said deformity,
* have reached or are over 65 years of age,
* present with normal or corrected vision,
* capable of walking independently without the use of an assistive device, since the use of technical aids masks the potential effects of the insole.

Exclusion Criteria:

* present with a current injury, or injury 6 months prior to the test, in the lower limb,
* Suffer from a musculoskeletal disorder,
* present with uncorrected vision,
* are pregnant,
* experience neurological disorders, diabetes or lower limb amputation/prosthetics, plantar ulcers, or cognitive impairment

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Stabilometry | Pre intervention, 3 months post intervention, 6 months post intervention
  To evaluate balance, participants were instructed to maintain the protocol anthropometric position proposed by the International Society for the Advancement of Kinanthropometry (ISAK); participants positioned their head on the Frankfort plane, with their upper limbs in a relaxed position, palms facing forward, and thumbs separated from the rest of their fingers.
  Participants were required to stand barefoot, with feet externally rotated at 30 degrees and a distance of 4 cm between both heels.
  A Gyko inertial sensor system was used to collect the balance data (i.e. ellipse area (EA): length and surface area in cm2). The software automatically calculates the length and surface projection, the velocity projection and the frequency of oscillations. The Gyko system offers high reliability in measuring postural control compared to other measurement systems . Previous research has shown that this protocol had moderate to strong evidence of validity and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernández de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hertel J, Sloss BR, Earl JE. Effect of foot orthotics on quadriceps and gluteus medius electromyographic activity during selected exercises. Arch Phys Med Rehabil. 2005 Jan;86(1):26-30. doi: 10.1016/j.apmr.2004.03.029. PMID 15640985
- [Result] Hatton AL, Dixon J, Martin D, Rome K. The effect of textured surfaces on postural stability and lower limb muscle activity. J Electromyogr Kinesiol. 2009 Oct;19(5):957-64. doi: 10.1016/j.jelekin.2008.04.012. Epub 2008 Jun 18. PMID 18565764
- [Result] Kulig K, Burnfield JM, Reischl S, Requejo SM, Blanco CE, Thordarson DB. Effect of foot orthoses on tibialis posterior activation in persons with pes planus. Med Sci Sports Exerc. 2005 Jan;37(1):24-9. doi: 10.1249/01.mss.0000150073.30017.46. PMID 15632663